CLINICAL TRIAL: NCT06982040
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of NTQ5082 Capsules in the Treatment of Patients With Primary IgA Nephropathy
Brief Title: Evaluate the Efficacy and Safety of NTQ5082 Capsules in Patients With Primary IgA Nephropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTQ5082-202
Record Dates: First submitted 2025-05-12; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NTQ5082 capsules 100 mg (Experimental): NTQ5082 capsules 100 mg
  Interventions: Drug: NTQ5082 capsules 100 mg
- NTQ5082 capsules 200 mg (Experimental): NTQ5082 capsules 200 mg
  Interventions: Drug: NTQ5082 capsules 200 mg
- NTQ5082 capsules 300 mg (Experimental): NTQ5082 capsules 300 mg
  Interventions: Drug: NTQ5082 capsules 300 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTQ5082 capsules 100 mg — NTQ5082 capsules 100 mg
  Arms: NTQ5082 capsules 100 mg
Drug: NTQ5082 capsules 200 mg — NTQ5082 capsules 200 mg
  Arms: NTQ5082 capsules 200 mg
Drug: NTQ5082 capsules 300 mg — NTQ5082 capsules 300 mg
  Arms: NTQ5082 capsules 300 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
NTQ5082 is a small molecule inhibitor of complement factor B (CFB) that inhibits the enzymatic activity of CFB, thereby blocking the alternative pathway of the complement activation cascade. It is being clinically developed for the treatment of primary IgA nephropathy The main objectives of the study were to assess the efficacy and safety of NTQ5082 capsules in the treatment of patients with primary IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female.
2. Body weight ≥40 kg, BMI between 15 to 38 kg/m².
3. Diagnosis of primary IgA nephropathy confirmed by renal biopsy within 8 years before screening or during screening.
4. 24-hour urine protein excretion (24h-UPE) ≥0.75 g/24h, or first morning void (FMV) urine protein-to-creatinine ratio (UPCR) ≥0.8 g/g.
5. Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73m².
6. Previously vaccinated with ACYW135 meningococcal polysaccharide vaccine and pneumococcal vaccine.
7. Received renin-angiotensin system (RAS) inhibitor therapy for at least 12 weeks prior to randomization, with stable treatment at the maximum recommended dose or maximum tolerated dose of RAS inhibitors for at least 4 weeks prior to randomization.
8. Agreement to use at least one effective contraceptive method with partners during sexual activity from signing the informed consent form until 4 weeks after the last administration of the investigational product, and refrain from sperm/egg donation during this period.

Exclusion Criteria:

1. Receipt of aldosterone receptor antagonists, renin inhibitors, or medications significantly affecting creatinine levels within 4 weeks or 5 half-lives (whichever is longer) before first investigational product administration.
2. Continuous use of systemic corticosteroids, immunosuppressants/modulators, or Chinese herbal medicines with immunosuppressive effects within 12 weeks or 5 half-lives (whichever is longer) before first investigational product administration.
3. Treatment with biological agents or complement pathway inhibitors (other than the study drug) within 12 weeks or 5 half-lives (whichever is longer) before first investigational product administration.
4. History of gastrointestinal surgery potentially altering drug absorption/distribution/metabolism/excretion, severe gastrointestinal disorders, or conditions causing dysphagia/recurrent vomiting that may interfere with oral medication intake.
5. Major trauma/surgery within 12 weeks before screening or planned major surgery during the study.
6. Previous bone marrow/hematopoietic stem cell transplantation or solid organ transplantation (e.g., heart, lung, kidney, liver).
7. Known/suspected hereditary complement deficiency, or diagnosed primary/severe secondary immunodeficiency.
8. Poorly controlled blood pressure as assessed by the investigator.
9. Poorly controlled blood glucose as assessed by the investigator.
10. Presence of nephrotic syndrome, rapidly progressive glomerulonephritis, renal pathology showing >50% glomerular crescents, or >50% tubular atrophy-interstitial fibrosis.
11. Participation in other interventional clinical trials with pharmacological/device interventions within 4 weeks before screening.
12. Pregnant/lactating women or those planning pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The log-transformed ratio of 24-hour urine protein-to-creatinine ratio (24h-UPCR) compared to baseline after 12 weeks of treatment. | Week 12

SECONDARY OUTCOMES:
The log-transformed ratio of 24-hour urine protein-to-creatinine ratio (24h-UPCR) compared to baseline during treatment period except week 12 | From week 1 to week 24
The change in estimated glomerular filtration rate(eGFR) compared to baseline during treatment period. | From week 1 to week 24
The change in serum creatinine (SCr) compared to baseline during treatment period. | From week 1 to week 24
The log-transformed ratios of first morning void (FMV) UPCR and UACR compared to baseline during treatment period | From week 1 to week 24
The change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale score compared to baseline during the treatment period. | From week 1 to week 24
  0-52,the higher the score, the better the QOL.
Incidence and severity of adverse events [safety and tolerability] | 28weeks
  Adverse events were based on clinically significant laboratory tests, vital signs, physical examination, and 12-lead electrocardiography